CLINICAL TRIAL: NCT00588263
Title: Anonymous Testing of Pathology Specimens for BRCA Mutations in Ashkenazi Jewish Individual With Cancer
Brief Title: Anonymous Testing of Pathology Specimens for BRCA Mutations in Ashkenazi Jewish Individuals Who Have Cancer
Status: Withdrawn | Type: Observational
Why Stopped: Data from MSK-IMPACT is sufficient for relevant analyses going forward
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 00-087
Record Dates: First submitted 2007-12-22; First posted 2008-01-08 (Estimated); Last update posted 2018-02-19 (Actual); Status verified 2017-08

CONDITIONS: Extrahepatic Bile Duct Cancer; Gallbladder Cancer; Gastric Cancer; Lung Cancer; Melanoma; Non-Hodgkin's Lymphoma; Uterine Cancer; CORPUS UTERI,ENDOMETRIUM; LUNG; OVARY
Keywords: Ashkenazi Jewish; Cancer; 00-087
MeSH Terms: conditions — Bile Duct Neoplasms; Gallbladder Neoplasms; Stomach Neoplasms; Lung Neoplasms; Melanoma; Lymphoma, Non-Hodgkin; Uterine Neoplasms; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blocks or extracted DNA from patients who have identified themselves as Jewish will be obtained and a determination will be made as to whether there is adequate material to proceed without exhausting the block or extracted DNA.
  Four unstained sections (research specimens) or paraffin "curls" will be cut from each block. In those cases where a block containing normal resection margin or any other biopsy of normal tissue are available, tissue will be cut from this block so as to preserve tumor tissue for later investigators. It is not necessary for sections to be reviewed to confirm that tumor is present in the section, since any germline DNA is adequate for this analysis.
Oversight: Data Monitoring Committee: No

SUMMARY:
The intent of the proposed study is to describe the prevalence of the most common recurring mutations in BRCA1 and BRCA2, blmAsh , and the A636P MSH2 mutation among Ashkenazi Jewish individuals with a variety of cancer diagnoses. If a substantial proportion of these samples contain such mutations, future patients presenting with these diseases may wish to undergo genetic counseling and, if appropriate, formal genetic testing. The benefit from such a process would pertain mainly to the families of these individuals.

DETAILED DESCRIPTION:
Germline mutations in the genes BRCA1 and BRCA2 have been demonstrated in the majority of hereditary breast and ovarian cancer families. The increased risk to develop both breast and ovarian cancer associated with inheriting a BRCA1 or BRCA2 mutation has been well established. It has also been suggested that is an overrepresentation of other cancers such as colon, prostate and pancreatic cancer present in BRCA1 or BRCA2 families. Population specific mutations in BRCA1 and BRCA2 have been identified. In the Ashkenazi Jewish population, 3 specific mutations have been seen in 2% of the population. This study will anonymously screen archived tissue samples of Ashkenazi Jewish individuals diagnosed with cancer between 1993 and 1996 at MSKCC for the three founder mutations seen in the Ashkenazi Jewish population. Results will be stratified by tumor type and compared with the population frequency to determine whether individuals inheriting mutations in BRCA1 or BRCA2 may have an increased risk to develop other cancers, in addition to breast and ovarian cancer. This information will be useful in helping to identify individuals who may benefit from genetic counseling and possibly genetic testing who to date are not typically referred. It will also be useful in developing high-risk cancer screening strategies and determining appropriate options for prophylactic surgery.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of cancer made at MSKCC or collaborating institutions, AND
* Tissue block of tumor or normal margin or extracted DNA available for study and sufficient material present to allow study without exhausting block or DNA,
* Individual self-identified as Jewish on intake.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Cases will be identified in one of two ways. Pathology records will be reviewed for the years 1985-present. All patients with diagnoses of pancreatic cancer, uterine cancer,lymphoma, melanoma, cancer of the gallbladder and bile duct, stomach cancer, brain cancer, ovarian cancer, colon cancer, head and neck cancer, lung cancer and breast cancer(including DCIS) from 1985 to the present at MSKCC will be identified.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2000-07; Primary Completion 2018-07 (Estimated); Study Completion 2018-07 (Estimated)

PRIMARY OUTCOMES:
determine the prevalence of recurring BRCA1 and BRCA2 mutations | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Offit, M.D., Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org